CLINICAL TRIAL: NCT04946578
Title: Modulation of the Intestinal Microbiome, and Its Effects on Endurance Exercise Capacity in Moderately Trained Individuals
Brief Title: The Effect of Prebiotics on Endurance Performance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University (Other)
Responsible Party: Principal Investigator, Fred Troost, Principal Investigator, Maastricht University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sport and microbiota
Record Dates: First submitted 2021-05-05; First posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Microtia
MeSH Terms: conditions — Congenital Microtia | interventions — Prebiotics

STUDY DESIGN:
Intervention Model Description: The study conforms to a randomized, single-blinded, placebo-controlled parallel study design.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prebiotic intervention group (Experimental): Prebiotic supplementation
  Interventions: Dietary Supplement: Prebiotic
- Placebo control group (Placebo Comparator): Maltodextrin
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Prebiotic — 6 weeks of prebiotic supplementation twice a day
  Arms: Prebiotic intervention group
Other: Placebo — 6 weeks of maltodextrin supplementation twice a day
  Arms: Placebo control group

SUMMARY:
The aim of this study is to investigate the effect of a six-week period personalised food intervention with prebiotic supplementation on intense exercise performance in healthy, recreationally active adults.

DETAILED DESCRIPTION:
The study conforms to a randomized, single-blinded, placebo-controlled parallel study design.

a prebiotic supplement will be selected based on a participants gut microbiota. 1 sachet of prebiotic or placebo will be given twice a day over a period of 6 weeks.

Before the start of the study, a VO2max test will be performed. Subjects will bring faecal samples which is collected at home. A time to exhaustion of approximately 80% of their VO2max will be performed at baseline and after the 6 weeks intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 - 40 y
* BMI range 18.5 - 25 kg/m2
* Recreational active (performing non-competitive physical endurance exercise at least two times per week with a minimum duration of 60 minutes per exercise bout)

Exclusion Criteria:

* Smoking
* Performing regular resistance training (3+ times per week, carrying out progressive overload training)
* Subject following an overly imbalanced or restrictive diet as per nutritional advice
* Participants who received antibiotics in the 90 days prior to the start of the study
* Self-admitted lactose intolerance
* Administration of probiotic or prebiotic supplements in the 14 days prior to the study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2020-08-24 (Actual); Primary Completion 2021-08-23 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Time to Exhaustion | From baseline to end of the study (up to max 45 days)
  Time on cycle ergometer until exhaustion

SECONDARY OUTCOMES:
Gut microbiota composition | From baseline to end of the study (up to max 45 days)
  Composition of the gut microbiota by faecal sample analysis
Plasma short chain fatty acids | From baseline to end of the study (up to max 45 days)
  Short chain fatty acids in plasma
Blood glucose | From baseline to end of the study (up to max 45 days)
  Fasted blood glucose
Insulin | From baseline to end of the study (up to max 45 days)
  Fasted insulin
Intestinal permeability by sugar test | From baseline to end of the study (up to max 45 days)
  Intestinal permeability measured by a sugar drink test

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No